CLINICAL TRIAL: NCT04174846
Title: Comparison of Treatment of Severe Acute Malnutrition in Children 6-59 Months Old With Ready-to-use Therapeutic Food and Ready-to-use-supplementary Food: An Individual Randomized, Double-Blind, Controlled, Clinical Non-Inferiority Trial
Brief Title: Comparison of Treatment of SAM in Children 6-59 Months With RUTF and RUSF in Umerkot, Sindh, Pakistan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19
Sponsor: Aga Khan University (Other)
Collaborators: United Nations World Food Programme (WFP) (Other); People's Primary Healthcare Initiative (PPHI), Sindh (Unknown)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Professor & Associate Director, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-1615-4895
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of SAM children with RUTF (Active Comparator): Treatment of severe acute malnutrition (SAM) in children 6-59 months old with standard ready-to-use therapeutic food (RUTF)
  Interventions: Dietary Supplement: Ready-to-use therapeutic food (RUTF)
- Treatment of SAM children with RUSF (Experimental): Treatment of severe acute malnutrition (SAM) in children 6-59 months old with ready-to-use-supplementary food (RUSF)
  Interventions: Dietary Supplement: Ready-to-use-supplementary food (RUSF)

INTERVENTIONS:
Dietary Supplement: Ready-to-use therapeutic food (RUTF) — SAM children will receive approximately 190 kcal/kg/day of standard RUTF
  Arms: Treatment of SAM children with RUTF
Dietary Supplement: Ready-to-use-supplementary food (RUSF) — SAM children will receive approximately 190 kcal/kg/day of Acha Mum (AM-RUSF)
  Arms: Treatment of SAM children with RUSF

SUMMARY:
In Pakistan, around 15% of children under five are wasted, which is almost twice that of the global prevalence 7.5%. There is a demand for a reliable and consistent locally available severe acute malnutrition (SAM) treatment option since currently the only option is to use an imported ready-to-use-therapeutic food (RUTF). While imported RUTF is successful for treatment of children with SAM, Pakistan is often faced with supply chain issues and consequentially management of SAM with RUTF is unreliable. The World Food Programme (WFP)'s work in Pakistan supports government-led efforts to improve food and nutrition security, including the development of Acha Mum, a chickpea containing lipid-based ready-to-use-food. Acha Mum replaces the peanut in standard RUTF formulation with chickpea, a locally available legume. Acha Mum is well accepted by children in Pakistan and is currently being used as a treatment for children with moderate acute malnutrition (MAM) in targeted supplementary feeding programs (TSFP) throughout the country. The broad objective of this clinical trial is to test the effectiveness of a chickpea-based specialized nutritious food Acha Mum, compared to a standard RUTF for the treatment of SAM. The study will be conducted in 10 basic health units (BHUs) operating by PPHI in Umerkot district of Sindh, Pakistan. This will be an individual randomized, double-blinded, controlled clinical non-inferiority trial assessing the treatment of SAM with one of two therapeutic foods. A total of 1700 children will be part of the study (850 children in RUTF and 850 children in Acha Mum group). Children aged 6-59 months with SAM, i.e. MUAC <11.5 cm and/or with bilateral pitting oedema (+, ++), with appetite and without medical complications presenting at selected rural therapeutic feeding clinics. The primary outcome is recovery from SAM, deﬁned as: MUAC ≥ 11.5cm (for two consecutive weekly visits), clinically well, no bilateral pitting oedema (for two consecutive weekly visits). The secondary outcomes include neurocognitive performance after first 4 weeks of treatment as assessed by eye tracking and infant problem solving; changes in MUAC, weight, and length; time to recovery from SAM; time to recovery from MAM defined as achieved a MUAC ≥12.5 cm; relapse into MAM; relapse into SAM and any adverse events.

DETAILED DESCRIPTION:
Rationale: In Pakistan, around 15% of children under five are wasted, which is almost twice that of the global prevalence 7.5%. There is a demand for a reliable and consistent locally available severe acute malnutrition (SAM) treatment option since currently the only option is to use an imported ready-to-use-therapeutic food (RUTF). While imported RUTF is successful for treatment of children with SAM, Pakistan is often faced with supply chain issues and consequentially management of SAM with RUTF is unreliable. The World Food Programme (WFP)'s work in Pakistan supports government-led efforts to improve food and nutrition security, including the development of Acha Mum, a chickpea containing lipid-based ready-to-use-food. Acha Mum replaces the peanut in standard RUTF formulation with chickpea, a locally available legume. Acha Mum is well accepted by children in Pakistan and is currently being used as a treatment for children with moderate acute malnutrition (MAM) in targeted supplementary feeding programs (TSFP) throughout the country.

Objectives: The broad objective of this clinical trial is to test the effectiveness of a chickpea-based specialized nutritious food Acha Mum, compared to a standard RUTF for the treatment of SAM.

Study Area: The study will be conducted in 10 basic health units (BHUs) operating by PPHI in Umerkot district of Sindh, Pakistan.

Study Design: This will be an individual randomized, double-blinded, controlled clinical non-inferiority trial assessing the treatment of SAM with one of two therapeutic foods.

Sample Size: A total of 1700 children will be part of the study (850 children in RUTF and 850 children in Acha Mum group).

Study Population: Children aged 6-59 months with SAM, i.e. MUAC <11.5 cm and/or with bilateral pitting oedema (+, ++), with appetite and without medical complications presenting at selected rural therapeutic feeding clinics.

Timeline: The duration of study will be 24 months (3 months for protocol and tool development, 18 months for enrollment and follow-ups and 3 months for data cleaning, analysis and report writing.

Expected outcomes: The primary outcome is recovery from SAM, deﬁned as: MUAC ≥ 11.5cm (for two consecutive weekly visits), clinically well, no bilateral pitting oedema (for two consecutive weekly visits). The secondary outcomes include neurocognitive performance after first 4 weeks of treatment as assessed by eye tracking and infant problem solving; changes in MUAC, weight, and length; time to recovery from SAM; time to recovery from MAM defined as achieved a MUAC ≥12.5 cm; relapse into MAM; relapse into SAM and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-59 months with SAM, i.e. MUAC <11.5 cm
* Bilateral pitting oedema (+,++)
* Appetite
* Without medical complications

Exclusion Criteria:

* Children will be excluded if they were simultaneously involved in another research trial or supplemental feeding program
* Developmentally delayed
* Have a chronic debilitating illness such as cerebral palsy (not including HIV or TB)
* Had a history of milk or peanut allergy.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Recovery rate from SAM | 12 weeks
  Number of children recovered from SAM, deﬁned as: MUAC ≥ 11.5cm (for two consecutive weekly visits), clinically well, no bilateral pitting oedema (for two consecutive weekly visits)

SECONDARY OUTCOMES:
Neurocognitive performance after first 4 weeks of treatment | 4 weeks
  Neurocognitive performance after first 4 weeks of treatment as assessed by eye tracking and infant problem solving
Changes in mid-upper arm circumference (MUAC) | 12 weeks
  Changes in MUAC will be assessed by cm & mm
Changes in weight | 12 weeks
  Changes in weight will be assessed by grams
Changes in length | 12 weeks
  Changes in length will be assessed by cm
Time to recovery from SAM | 12 weeks
  Time to recovery from MAM defined as achieved a MUAC ≥12.5 cm
Relapse rate into SAM | 24 weeks
  Number of relapse in SAM will be identified after 3 months of follow-up
Non-responder children | 12 weeks
  Number of children who non-responded will be assessed in follow-up visits
Defaulter children | 24 weeks
  Number of defaulter children during the study will be assessed by follow-up visits
Adverse events | 24 weeks
  Number of adverse events (if any) will be identified in follow-up visits

CONTACTS AND LOCATIONS:
Locations (1):
- 10 Basic Health Units (BHUs) operating by People's Primary Healthcare Initiative (PPHI), Umarkot, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared